CLINICAL TRIAL: NCT06047860
Title: A Clinical Study of Recombinant Human Vascular Endothelial Inhibitor (Endo) in Combination With Bragg Treatment for Advanced Refractory Non-small Cell Lung Cancer
Brief Title: A Clinical Study of Recombinant Human Vascular Endothelial Inhibitor in Combination With PRaG for Advanced Refractory Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2022-173-01
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor; Refractory Tumor
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy; Immune Checkpoint Inhibitors; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): M-CSF 200 μg administered subcutaneously daily for 7 days on the first day of treatment; IL-2 2 million IU administered subcutaneously daily for 7 days the day after GM-CSF; PD-1/PD-L1 inhibitor within one week of radiotherapy; Recombinant human vascular endothelial inhibitor (Endo) 210 mg CIV72h starting on the first day of treatment, every 21 days for a minimum of ≥ 2 cycles of this combination therapy.
  Maintenance treatment phase:
  Maintenance with PD-1/PD-L1 inhibitor in combination with recombinant human vascular endothelial inhibitor (Endo) until progression or intolerable side effects.
  Interventions: Radiation: Radiotherapy; Drug: PD-1/PD-L1 inhibitor; Drug: Granulocyte-macrophage colony-stimulating factor subcutaneous injection; Drug: Interleukin 2 subcutaneous injection; Drug: Endostatin

INTERVENTIONS:
Radiation: Radiotherapy — hypofractionated radiotherapy/SBRT
  Other Names: SBRT
Drug: PD-1/PD-L1 inhibitor — PD-1/PD-L1 inhibitor within one week of radiotherapy
  Other Names: PD-1/PD-L1 antibody
Drug: Granulocyte-macrophage colony-stimulating factor subcutaneous injection — IL-2 2 million IU the day after the end of GM-CSF, administered subcutaneously daily for 7 days;
  Other Names: GM-CSF
Drug: Interleukin 2 subcutaneous injection — IL-2 2 million IU the day after the end of GM-CSF, administered subcutaneously daily for 7 days;
  Other Names: IL-2
Drug: Endostatin — Recombinant human vascular endothelial inhibitor (Endo) 210 mg CIV72h was started on the first day of treatment, every 21 days for a minimum of ≥ 2 cycles of this combination therapy.
  Other Names: Endo

SUMMARY:
Exploring the efficacy and safety of recombinant human vascular endothelial inhibitor (Endo) in combination with Bragg therapy in advanced refractory non-small cell lung

DETAILED DESCRIPTION:
Radiotherapy:

Start radiotherapy on the first day of treatment, as described in 6.2 above;

GM-CSF treatment:

GM-CSF 200 μg on the first day of treatment, administered subcutaneously daily for 7 days; IL-2 treatment. 2 million IU of IL-2 on the day after GM-CSF, administered subcutaneously daily for 7 days;

Immunotherapy:

PD-1/PD-L1 inhibitors within one week of radiotherapy;

Recombinant human vascular endothelial inhibitor (Endo):

Recombinant human vascular endothelial inhibitor (Endo) 210 mg CIV72h starting on the first day of treatment, every 21 days for a minimum of ≥ 2 cycles of this combination therapy.

Maintenance treatment phase:

Maintenance with PD-1/PD-L1 inhibitor in combination with recombinant human vascular endothelial inhibitor (Endo) until progression or intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years;
2. Patients enrolled must be eligible for patients with recurrent or metastatic advanced non-small cell lung cancer, with a clear pathological diagnosis report or history of disease, with guidelines that do not clearly recommend standard treatment regimens or who are unable to tolerate standard treatment regimens, and with clear measurable metastatic lesions (>1cm);
3. No congestive heart failure, unstable angina, or unstable arrhythmia within the last 6 months.
4. Patient activity status score of 0-3 on the Eastern Cooperative Oncology Group (ECOG) scale with life expectancy assessed at ≥3 months.
5. No previous severe haematopoietic, cardiac, pulmonary, hepatic or renal abnormalities and immunodeficiency.
6. Absolute T-lymphocyte values ≥ 0.5 times the lower limit of normal and neutrophils ≥ 1.0 x 109/L; AST and ALT ≤ 3.0 times the upper limit of normal (≤ 5.0 times the upper limit of normal for hepatocellular carcinoma/metastatic liver cancer); creatinine ≤ 3.0 times the upper limit of normal, 1 week prior to enrollment.
7. Patients must have the ability to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. Persons with a history of other malignant disease in the last 5 years, except cured skin cancer and carcinoma in situ of the cervix;
3. Persons with a history of uncontrolled epilepsy, central nervous system disorders or psychiatric disorders whose clinical severity, as judged by the investigator, may prevent the signing of an informed consent or affect the patient's compliance with drug therapy;
4. Clinically significant (i.e., active) cardiac disease such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmias requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months;
5. Persons requiring immunosuppressive therapy for organ transplantation;
6. Known major active infection or, in the judgement of the investigator, major haematological, renal, metabolic, gastrointestinal, endocrine dysfunction or metabolic disorders, or other serious uncontrolled concomitant disease;
7. Hypersensitivity to any investigational drug component;
8. Persons with a history of immunodeficiency, including those who have tested positive for HIV or have other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, or other immune-related diseases requiring long-term oral hormone therapy
9. Persons with active tuberculosis infection;
10. Those with interstitial lung disease or non-infectious pneumonia that may prevent the assessment of pulmonary toxicity associated with the study or the manager;
11. Other conditions that, in the opinion of the investigator, are not suitable for enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate(ORR) | six weeks
  ORR is defined as the proportion of patients who have a partial (PR) or complete response (CR) to therapy among the total number of evaluable patients.
Disease control rate (DCR) | six weeks
  the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD)
Progression free survival (PFS) | six weeks
  The time from commencement of treatment to disease progression or death from any cause.
Overall survival (OS) | six weeks
  The time from the first day of enrollment to death from any cause.
Incidence of adverse events | six weeks
  the rate of AE

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of SchoowUniversity, Suzhou, China

IPD SHARING:
Plan to Share IPD: No